CLINICAL TRIAL: NCT05988060
Title: The Effect of Physical Exercise During Radiotherapy on Physical Functioning in Patients With Head and Neck Cancer: a Trial Within Cohorts, the VITAL Study
Brief Title: Physical Exercise for Patients With Head and Neck Cancer
Acronym: VITAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Verbeeten (Other)
Collaborators: Verbeeten Fonds (Unknown); Stichting Fight Cancer (Unknown); CZ Fonds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL79549.028.21
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; chemo- or bioradiotherapy; physical exercise intervention; physical performance; trial within cohorts; TwiCs
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study a TwiCs design will be used. The TwiCs design consists of an experimental intervention study within an observational longitudinal cohort. This design uses a staged-informed consent. Patients will be asked to participate in an observational longitudinal cohort study and will be informed about the design with the probability to be randomly invited for an experimental intervention which they can accept or refuse. When patients are willing to participate in the observational longitudinal cohort, an informed consent (IC) will be signed. Directly after cohort enrollment, all patients will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who were randomized in the PEI group and accepted the invitation (Experimental): The experimental intervention consist of a PEI for 10 weeks. The PEI will be executed 6 to 7 weeks during and 3 to 4 weeks after (C/B)RT.
  Interventions: Other: Experimental Intervention
- Patients who were not randomized in the PEI group (No Intervention): Patients will receive usual care.

INTERVENTIONS:
Other: Experimental Intervention — Patients who were randomized in the PEI group and accepted the invitation to undergo the experimental intervention receive a PEI for 10 weeks. The PEI will be executed 6 to 7 weeks during and 3 to 4 weeks after (C/B)RT. The PEI consists of a 60 minutes intervention twice a week and will be supervised by a physiotherapist specialized in oncology.
  Patients who receive the intervention also have to do home-based aerobic and muscle strength exercises by themselves three times a week.
  Other Names: Physical Exercise Intervention
  Arms: Patients who were randomized in the PEI group and accepted the invitation

SUMMARY:
The goal of this trial within cohorts study is to determine and compare physical performance, muscle strength, fatigue, quality of life, body composition, nutritional status, physical activity, treatment tolerability of radiotherapy (RT), chemoradiation (CRT) or bioradiation (BRT), and healthcare related costs in patients with head and neck cancer (HNC) with and without a 10 week physical exercise intervention (PEI) during RT, CRT or BRT ((C/B)RT).

Patients who were randomized in the PEI group and accepted the invitation to undergo the experimental intervention receive a PEI twice a week for 10 weeks. The PEI will be executed 6 to 7 weeks during and 3 to 4 weeks after (C/B)RT.

Researchers will compare patients who undergo the PEI with patients who did not undergo the PEI to see if there is difference in physical performance, muscle strength, fatigue, Quality of Life, body composition, nutritional status, physical activity, treatment tolerability of (C/B)RT , and healthcare related costs in patients with Head and Neck Cancer (HNC) with and without a 10 week Physical Exercise Intervention (PEI) during (C/B)RT).

ELIGIBILITY:
Inclusion Criteria:

1. patients with HNC who are scheduled for (C/B)RT,
2. ≥18 years of age,
3. sufficient Dutch writing and reading skills,
4. a Karnofsky performance status (KPS) >60,
5. able to walk ≥60m without a mobility aid, and
6. no contraindication for physical activity as measured with the physical activity readiness questionnaire (PAR-Q).

Exclusion Criteria:

1. recurrence of HNC and/or
2. secondary HNC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-11-09 (Estimated); Study Completion 2026-11-09 (Estimated)

PRIMARY OUTCOMES:
physical performance | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  six minute walking test

SECONDARY OUTCOMES:
Muscle strength | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Grip strength
Muscle strength | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  30 seconds chair to stand test
Muscle strength | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Microfet handheld dynamometer
Health Related Quality of Life | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Assessed by the EuroQol- five dimensions- five level (EQ-5D-5L). This questionnaire contains 6 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and a total score for global health. The first 5 item have 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The score of these item can range from 0 to 4. The higher the total score of these five items, the lower the quality of live. The global health scores on a range 0-100. The higher the score of this item, the higher the global health.
Health Related Quality of Life | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Assessed by the European organisation for research and treatment for cancer quality of life questionnaire (EORTC QLQ-C30). This questionnaire contains 30 questions scoring 9 subscales and 6 single items: 5 functional scales, 3 symptom scales and 1 global health / quality of life scale. The score of each subscale of single items ranges from 0 to 100. A higher score on the functional scales means a high level of functioning. A higher score on the symptom scales means a high level of experiencing symptoms. A higher score on global health / quality of life means a high score of quality of life.
Health Related Quality of Life | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Assessed by the European organisation for research and treatment for cancer quality of life questionnaire head and neck module (EORTC-QLQ-H&N43). This questionnaire contains 43 specific head and neck cancer questions scoring 19 subscales of symptoms. The higher the score of the subscale, the higher the level symptomology.
Fatigue | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Assessed by the multidimensional fatigue inventory (MFI). The MFI contains 20 items scoring the following domains: general, physical and mental fatigue, and reduced activity and motivation. Every scale scores 4 till 20. The greater the score, the more fatigue or limitations in live because of fatigue.
Body composition | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  body mass index (BMI)
Nutrition status | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Assessed by the short nutritional assessment questionnaire (SNAQ). The short nutritional assessment questionnaire (SNAQ) consists of three questions and will be used to monitor nutritional status and assess the risk of malnutrition. The total score of this questionnaire ranges from 0 to 7. 0 means no nutritional problems and a high score means malnutrition.
Physical activity | M0 (baseline/before (C/B)RT), M1 (12 weeks), M2 (6 months), M3 (12 months)
  Assessed by the short questionnaire to assess health enhancing physical activity (SQUASH). The SQUASH measures the frequency, duration and intensity of 4 different physical activity: physical activity going to work, physical activity during household activity, physical activity at work, physical activity in spare time. The higher the score, the higher the level of physical activity.
Tolerability of radiotherapy, chemoradiation or bioradiation | M1 (12 weeks), M2 (6 months), M3 (12 months)
  tolerability will be retrieved from medical records and registered as the percentage of scheduled treatment completion, percentage of (C/B)RT adjustment and type of (C/B)RT adjustment.
socio-demographic data and medical data | M0 (baseline/before (C/B)RT)
  age, gender, education, employment, marital status tumour site, disease stage, comorbidity, HPV status, tobacco and alcohol use, nutrition status and type of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Kriellaars, Msc., Principal Investigator — Instituut Verbeeten
Locations (1):
- Instituut Verbeeten, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kriellaars Y, Vermaire JA, Beugeling M, Poorter R, Drijvers J, Speksnijder CM. The effect of physical exercise during radiotherapy on physical performance in patients with head and neck cancer: a trial within cohorts study protocol, the vital study. BMC Cancer. 2024 Apr 1;24(1):403. doi: 10.1186/s12885-024-12172-2. PMID 38561708